CLINICAL TRIAL: NCT06801990
Title: The Effect of Needle Insertion Angle on Contrast Distribution and Treatment Outcomes in S1 Transforaminal Epidural Steroid Injections
Acronym: Transforaminal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAR.FTR.BAP.01; Marmara University (Other: Marmara University Ethics Committee)
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain (LBP); Lumbar Radiculopathy; Intravascular Injection
Keywords: lumbar radicular pain , epidural injection , intravascular injection , contrast spread pattern , low back pain
MeSH Terms: conditions — Low Back Pain; Radiculopathy | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oblique Angle Group (Active Comparator): After the optimal image is obtained by angling the C-arm fluoroscopy in the cranial direction, the fluoroscopy will also be angled ipsilaterally obliquely.
  Interventions: Procedure: S1 transforaminal epidural steroid(dexamethasone) injection
- Non-Oblique Angle Group (Active Comparator): In order to visualize the S1 foramen, the C-arm scope will be open towards the cranial direction in AP imaging and no oblique angle will be given. In this group of patients, the needle entry point will be determined after the angle is given towards the cranial direction and the foramen is visualized.
  Interventions: Procedure: S1 transforaminal epidural steroid(dexamethasone) injection

INTERVENTIONS:
Procedure: S1 transforaminal epidural steroid(dexamethasone) injection — The designed study will examine the effect of oblique entry angles on contrast distribution patterns and treatment outcomes. Therefore, it aims to compare the smallest and largest angles that can be achieved under co-axial imaging at the S1 foramen. For this purpose, patients will be divided into two groups through randomization using a computer program. In the first group, after angling cranially and visualizing the foramen, the needle entry point will be determined. In the second group, after achieving optimal imaging by cranially angling the C-arm fluoroscope, an additional ipsilateral oblique angle will be applied to the fluoroscope.
  In this context, Plastaras et al. reported that an angle of 5° ± 5° is the most suitable range for the S1 foramen. Additionally, another study examining dorsal and ventral S1 foramen via tomography images found that the average angle providing the widest view of the dorsal foramen was 26.6° ± 3°. In the current study, no oblique angle will be applied

SUMMARY:
Nerve compression due to lumbar disc herniation (lumbosacral radiculopathy) is a condition characterized by pain in the lower back and legs and restricted lumbar joint movement due to the compression of nerves emerging from the lumbar spine caused by the protrusion of the intervertebral disc. Back pain negatively impacts patients' quality of life and emotional well-being. Treatment approaches aim to alleviate pain, improve joint mobility, and restore functionality through the use of pain-relief medications (topical or oral), physical therapy methods, and rehabilitation programs that include exercises for range of motion, stretching, and strengthening. When these approaches prove insufficient, interventional procedures (injection therapy) or surgical interventions come to the forefront.

One of the proven interventional treatment methods for herniated disc disease is the transforaminal epidural steroid injection (TFESE), which involves the injection of cortisone around the compressed nerve due to the herniation and is frequently performed in our clinic. Transforaminal injections require imaging guidance and the use of contrast media to enhance the safety and effectiveness of the procedure. To visualize the S1 foramen, needle entry is performed using various angles under fluoroscopy guidance. This study will investigate the effect of the needle entry angle on the spread and pattern of contrast media, complications, and treatment outcomes in fluoroscopy-guided S1 transforaminal epidural steroid injections. The research aims to determine whether the needle entry angle influences the pattern of contrast spread and the treatment outcomes in S1 TFESE.

Based on the findings of this study, the goal is to refine the procedure for patients requiring injections at this level in the future, optimizing the technique and clinical outcomes. This will provide essential insights to practitioners, maximize the benefits for the patient group undergoing the procedure, and make a significant contribution to medical science. Detailed information regarding the planned injection therapy by your algology specialist will be provided, and written and verbal consent will be obtained through the "Epidural Steroid Injection Consent Form." Various scales and questionnaires will be administered at specific intervals-prior to the procedure, 1 hour after, 3 weeks after, and 3 months after-to evaluate pain levels, treatment response, and the impact on daily activities. The content of these evaluations will be explained in detail by your physician.

Temporary side effects related to the injection may include increased pain at the injection site, low blood pressure, dizziness, fainting, and allergic reactions, all of which can be managed with appropriate treatment. Although rare, severe side effects such as nerve damage, spinal cord injury, or stroke have been reported in some cases. However, adherence to the guidelines outlined in treatment protocols and the performance of the procedure by adequately trained and experienced physicians significantly reduce the likelihood of these serious side effects. This injection will be performed by an algology specialist with at least 10 years of experience in this field. All necessary precautions will be taken against potential side effects, and the performing team will provide immediate medical intervention in case of complications.

Approximately 66 volunteers will participate in this study, with each follow-up evaluation expected to take about 15 minutes. The identities of participants will remain confidential, and they have the right to withdraw from the study at any time by notifying the researchers. If deemed necessary by the researchers, participants may also be excluded from the study. If a participant declines to participate or is excluded from the study, their treatment will not be interrupted. Participants will not bear any financial responsibility for research-related expenses, and no additional travel costs will be incurred as evaluations will coincide with regular clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Having S1 nerve root compression due to paravertebral disc herniation at the L5-S1 level detected by MRI
* Having history and physical examination findings consistent with S1 root compression
* Patients with low back and leg pain who have not responded to conservative treatment methods
* Being willing to participate in the study and having signed a consent form

Exclusion Criteria:

* Having undergone lumbosacral surgery
* Presence of transitional vertebra
* Presence of progressive motor deficit
* Presence of local and/or systemic infection
* History of malignancy
* Patients with lumbar disc herniation causing root compression outside the L5/S1 level on MRI
* Patients with bilateral S1 root compression on MRI
* Presence of spinal stenosis
* Pregnancy
* Presence of known coagulopathy
* Presence of known psychiatric disease diagnosis
* History of allergy to any of the injection materials
* Having received an epidural steroid injection within the last 3 months
* Receiving systemic steroid treatment for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
NRS | before intervention, 1 hour after intervention, 3 weeks after intervention, 3 months after intervention
  According to the Numeric Rating Scale (NRS): The Numeric Rating Scale is used to measure and monitor pain intensity. "0" represents no pain, and "10" represents the most severe pain imaginable. The patient rates their pain on a scale from 0 to 10. Due to its simplicity, this scale is frequently used in clinical research.
ODI | before intervention, 3 weeks after intervention, 3 months after intervention
  Oswestry Low Back Pain Disability Questionnaire (Oswestry Disability Index, ODI): It was developed to assess the degree of functional impairment in low back pain. It consists of 10 items. These items evaluate pain intensity, self-care, lifting-carrying, walking, sitting, standing, sleeping, the degree of pain variation, travel, and social life. Under each item, there are six statements from which the patient selects the one that best describes their condition. The first statement is scored as "0," and the sixth statement as "5." The total score is calculated, multiplied by two, and expressed as a percentage. The maximum score is "100," and the minimum score is "0." As the total score increases, the level of disability also increases.

SECONDARY OUTCOMES:
Contrast Spread Pattern | During the intervention
  Absence of anterior epidural spread will be considered stage 0, epidural spread at the needle entry level will be considered stage 1, and epidural spread detected in more than one segmental level will be considered stage 2. In addition, the staging system used by Jeong et al. will also be used. In this study, cephalic and caudal spread of contrast material in transforaminal injections were staged as follows: Grade 0, no visible spread; Grade 1, spread at the same vertebral level; Grade 2, spread at the level of upper intervertebral disc (IVD) (cephalic) or lower IVD (caudad); Grade 3 is defined as extension above the superior IVD, not exceeding the horizontal midline of the superior pedicle, or below the inferior IVD, not exceeding the horizontal midline of the inferior pedicle; Grade 4 is defined as extension above or below the horizontal midline of the superior or inferior pedicle, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara Üniversitesi Tıp Fakültesi, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No